CLINICAL TRIAL: NCT00829465
Title: Clinical Research of in the Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Clinical Research of Licartin Combined With TACE in the Treatment of Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-013
Record Dates: First submitted 2008-12-22; First posted 2009-01-27 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — metuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Active Comparator)
  Interventions: Procedure: Transcatheter arterial chemoembolization
- therapy (Experimental)
  Interventions: Drug: Licartin; Procedure: Transcatheter arterial chemoembolization

INTERVENTIONS:
Drug: Licartin — Licartin
  Other Names: TACE and Licartin
  Arms: therapy
Procedure: Transcatheter arterial chemoembolization — TACE

SUMMARY:
Liver cancer is a highly invasive malignancy and the rate of surgical resection is no more than 28%. After diagnosis, the average survival rate of patient is less than 50% in 6 month, less than 24% in 1 year and 5% in 5 year. The TACE treatment, under the theoretical basis of blood supply of Liver cancer, is obviously better than the other non-surgical therapy, in terms of tumor regression, AFP decrease, survival time and the evaluation of the quality of life. However, its overall effect is not yet satisfactory. As a result, concerning the research of drug for liver cancer and improving the overall efficacy of the treatment of liver cancer has a very real and important clinical significance and social value. Licartin (Iodine-131-Labeled Metuximab) injection is a antibody drug with new target and the only drug that China own the intellectual property rights. It has specific high affinity with HAb18G/CD147, the liver cell membrane antigen. Labeled 131I is taken to the liver tissue, owning high-dose concentration and releasing β particles to liver cancer cells to and kill cancer cells.

The Second Military Medical University, Eastern Hepatobiliary Surgery Hospital, planed to use the treatment of Licartin combined with TACE for the patients of unresectable hepatocellular carcinoma and evaluate the difference of tumor size, AFP change, TTP, the overall survival rate between different treatment group.

DETAILED DESCRIPTION:
Liver cancer is a highly invasive malignancy and the rate of surgical resection is no more than 28%. The TACE treatment, under the theoretical basis of blood supply of Liver cancer, is obviously better than the other non-surgical therapy, in terms of tumor regression, AFP decrease, survival time and the evaluation of the quality of life. Licartin injection is a antibody drug with new target and the only drug that China own the intellectual property rights. It has specific high affinity with HAb18G/CD147, the liver cell membrane antigen. Labeled 131I is taken to the liver tissue, owning high-dose concentration and releasing β particles to liver cancer cells to and kill cancer cells.

The Second Military Medical University, Eastern Hepatobiliary Surgery Hospital, planed to use the treatment of Licartin combined with TACE for the patients of unresectable hepatocellular carcinoma and evaluate the difference of tumor size, AFP change, TTP, the overall survival rate between different treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. the participation is entirely voluntary, good at compliance, sign the informed consent form in person;
2. diagnosed to be hepatocellular carcinoma by clinical method, imaging method and tumor markers; and the surgeons determine who can not undergo surgery;
3. confirmed to recurrent after surgery by pathology;
4. KPS score of physical state ≥ 60 points;
5. liver function is Child-Pugh A or B class

Exclusion Criteria:

1. General situation is poor and liver function Child-Pugh is C class;
2. there is a serious heart, kidney and blood system diseases in patients;
3. poor compliance;
4. there is allergy history of biological agents or in a state of allergy;
5. pregnancy and breast-feeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
OS of 1 years; TTP | 2008.12--2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Yang yefa, doctor, Study Director — Second Military Medical University